CLINICAL TRIAL: NCT02348749
Title: A Phase I/IIA Study of 18F-MFBG Imaging for Evaluation of Neuroendocrine Malignancies
Brief Title: 18F-MFBG Imaging for Evaluation of Neuroendocrine Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-138
Record Dates: First submitted 2015-01-19; First posted 2015-01-28 (Estimated); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Neuroendocrine Tumors
Keywords: 18F-MFBG Imaging; 14-138; PET/MR; PET/CT scan
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — 3-fluorobenzylguanidine; Positron-Emission Tomography; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: For phase I, a single dose of 18F-MFBG will be injected intravenously in patients. For all patients, pharmacokinetics and bio distribution will be evaluated using non invasive PET scanning and blood assays at multiple time points post injection. In the expansion phase, a single dose of 18F-MFBG will be injected intravenously followed by a single time point imaging using PET MR or PET/CT scanner

ARMS (1):
- pts with primary or metastatic neuroendocrine tumors (Experimental): For phase I, a single dose of 18F-MFBG will be injected intravenously in patients. For all patients, pharmacokinetics and bio distribution will be evaluated using non invasive PET scanning and blood assays at multiple time points post injection. In the expansion phase, a single dose of 18F-MFBG will be injected intravenously followed by a single time point imaging using PET MR scanner or PET/CT. In expansion cohort, an additional 50 patients with NB will be imaged. Patients will receive a single dose of 18F-MFBG intravenously, followed by a whole body PET scan on PET/CT or PET/CT scanner at 60-90 minutes post injection. Patients who show lesion detection by MFBG may be eligible for repeat imaging scan with 18 F- MFBG, at the discretion of PI or study investigator(s). All parameters and technical details of scanning will be as per the study and first imaging.
  Interventions: Radiation: 18F-MFBG (meta-fluoro benzylguanidine); Device: Positron emission tomography (PET) imaging; Other: Blood draws

INTERVENTIONS:
Radiation: 18F-MFBG (meta-fluoro benzylguanidine) — About 8mCi of 18F-MFBG will be administered to adult patients. Pediatric dose will be based upon adjustment using BSA to the dose of 8 mCi for 1.7m2 BSA ± 10% with maximum activity of 8 mCi. The tracer will be given intravenously.
Device: Positron emission tomography (PET) imaging — Dynamic imaging for the first 30 min over the chest and Whole body (WB) PET-CT scan. Imaging 2 (~1.0 - 2 hours post dose): Whole body (vertex to feet) PET-CT scan. Imaging 3 (~3-4 hours post dose): Whole body (vertex to feet) PET-CT scan.
Other: Blood draws — Blood samples to be collected: at baseline, 5, 15, 30, 60, 90, 120 and 180 mins post injection on the day of administration. (Phase I only)

SUMMARY:
The purpose of this study is to see how a new tracer named 18F-MFBG (Meta Fluorobenzyl Guanidine) behaves in the body after injection, how it spreads to all the organs and how it is removed from the body. We will also study how long 18F-MFBG lasts in the blood after administered. In addition we want to study if 18F-MFBG can show Neuroendocrine tumors on a PET-CT or PET MR scan.

ELIGIBILITY:
Inclusion Criteria:

Phase I:

* Eligible patients include patients with histologically proven Neuroendocrine tumors (paraganglioma, PHEO, or well differentiated NET of the lung or GI system) or NB. Patients who have NB, the diagnosis must be in accordance with the International Criteria, i.e., either histopathology or bone marrow involvement. Patients must be ≥5 years of age and able to undergo PET scan without sedation
* All patients must have MIBG-avid disease and evaluable disease on MIBG scan at the time of enrollment onto the protocol.
* Performance status of ≥60 on Karnofsky scale for patients >16 years of age and >60 on Lansky scale for patients <16 years of age.
* Cardiac, pulmonary, gastrointestinal and neurologic toxicity should all be ≤grade 2.

Expansion Cohort:

* Patients with diagnosis of NB (in accordance with the International Criteria, i.e., either histopathology or bone marrow involvement)
* Patients must be able to undergo PET scan without sedation
* Patients must have prior MIBG-avid disease and evaluable disease on MIBG scan at the time of enrollment onto the protocol.

  * If MIBG scan is available within 4 weeks of MFBG, with no intervening treatment, MIBG scan will not be repeated.
  * If prior MIBG scan is available >4 weeks of MFBG, MIBG scan will be done within a week (prior or after) of MFBG.
* Performance status of ≥60 on Karnofsky scale for patients >16 years of age and >60 on Lansky scale for patients ≤16 years of age.
* Cardiac, pulmonary, gastrointestinal and neurologic toxicity should all be ≤grade 2.
* Patients with positive lesion detection by 18F-MFBG may be eligible for repeat imaging scan, at the discretion of PI or study investigator(s).

Exclusion Criteria:

* Major organ toxicity including cardiac, pulmonary, gastrointestinal and neurologic toxicity more than grade 2.
* Active serious infections not controlled by antibiotics.
* Inability or unwillingness to undergo PET scanning
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Women who are pregnant or breastfeeding.
* Patient has an active malignancy of metastatic potential other than the known NE tumor for the past 3 years.
* Patients should not have received chemotherapy or radiation therapy (localized radiation therapy is allowed to non-evaluable sites) between prior 123I-MIBG scan and 18F-MFBG administration.
* Patients requiring anesthesia, who are not already undergoing anesthesia for standard-of-care procedures.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-03-17 (Actual)

PRIMARY OUTCOMES:
dosimetry of 18F MFBG | 1 year
  in two cohorts of patients: (a) those with NB and (b) those with non-NB NE. Data will be derived from blood draws and PET/CT scans at multiple time points after injection of 18F-MFBG IV.
radioactivity | 1 year
  Multiple samples will be counted and time activity curve generated for evaluation of serum clearance. Blood samples will be centrifuged and the plasma pipetted, weighed and counted to determine the plasma time activity concentration curves (% injected dose/liter), as well as for metabolite analysis of the 18F-MFBG compound by HPLC and/or TCA methodology.

SECONDARY OUTCOMES:
18 F-MFBG imaging PET/CT to target known sites of disease | 1 year
  Lesion detection will be evaluated based on per patient and per lesion basis. The segmental distribution method described for 123 I -MIBG imaging (modified curie scoring system will be used- appendix C). If, for each individual patient, there is a concordance of ≥70% of segments or lesion detection between MIBG and 18 F-MFBG , the latter will be considered as effectively targeting lesions. For discordant lesions, if MFBG imaging shows 2 or more lesions that are positive on other concurrent or follow up conventional imaging, it will be considered optimal targeting.

CONTACTS AND LOCATIONS:
Overall Officials: Neeta Pandit-Taskar, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/